CLINICAL TRIAL: NCT07101159
Title: Efficacy and Safety of Dalpiciclib Combined With Endocrine Adjuvant Therapy in Early-stage HR-positive/HER2-negative Breast Cancer: a Multicenter, Prospective Clinical Study
Brief Title: Dalpiciclib as Adjuvant Therapy for HR-positive/HER2-negative Early-stage Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-304
Record Dates: First submitted 2025-07-25; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Early Breast Cancer; Adjuvant Therapy; Hormone Receptor Positive / HER2-negative Breast Cancer
Keywords: dalpiciclib; hormone receptor positive/HER2-negative breast cancer; early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Tamoxifen; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-Year Dalpiciclib 125 mg + Endocrine Therapy (Experimental): Patients will receive dalpiciclib 125 mg orally once daily on days 1-21 of a 28-day cycle for 2 years, in combination with standard endocrine therapy.
  Interventions: Drug: Endocrine Therapy (Tamoxifen, Anastrozol, Letrozole, Exemestane); Drug: Dalpiciclib
- 3-Year Dalpiciclib 100 mg + Endocrine Therapy (Experimental): Patients will receive dalpiciclib 100 mg orally once daily on days 1-21 of a 28-day cycle for 3 years, in combination with standard endocrine therapy.
  Interventions: Drug: Dalpiciclib; Drug: Endocrine Therapy (Tamoxifen, Anastrozol, Letrozole, Exemestane)

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib 100 mg orally, daily on days 1-21 of a 28-day cycle, for 3 years.
  Arms: 3-Year Dalpiciclib 100 mg + Endocrine Therapy
Drug: Endocrine Therapy (Tamoxifen, Anastrozol, Letrozole, Exemestane) — Standard adjuvant endocrine therapy (e.g., tamoxifen or aromatase inhibitor), as per physician's choice.
Drug: Dalpiciclib — Dalpiciclib 125 mg orally, daily on days 1-21 of a 28-day cycle, for 2 years.
  Arms: 2-Year Dalpiciclib 125 mg + Endocrine Therapy

SUMMARY:
This study aims to evaluate the efficacy and safety of adjuvant endocrine therapy combined with dalpiciclib at different doses and durations in patients with hormone receptor (HR)-positive, HER2-negative early-stage breast cancer.

It is a multicenter, prospective clinical study. All enrolled patients will receive either dalpiciclib 125 mg for 2 years or dalpiciclib 100 mg for 3 years, in combination with standard endocrine therapy.

The primary endpoint is 3-year invasive disease-free survival (iDFS).

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients aged ≥ 18 years, who are postmenopausal or premenopausal/perimenopausal;
* Histologically confirmed HR-positive, HER2-negative early-stage breast cancer (immunohistochemical detection shows ER ≥ 10% and/or PR ≥ 10%, HER2 0-1+ or HER2 ++ but negative and non-amplified by FISH or CISH detection);
* Histologically confirmed invasive breast cancer with postoperative pathological stage II-III;
* Patients with or without prior neoadjuvant chemotherapy or adjuvant chemotherapy are eligible for enrollment;
* The maximum time from surgery to enrollment does not exceed 12 months;
* Patients receiving radiotherapy must have recovered from acute radiation reactions, with a washout period of at least 14 days from the end of radiotherapy to enrollment;
* Patients who received previous chemotherapy must have recovered from acute adverse reactions of chemotherapy (graded ≤ 1 according to [CTCAE]) before enrollment, except for alopecia or grade 2 peripheral neuropathy. There must be a washout period of at least 21 days from the last chemotherapy administration to enrollment;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* The main organ function levels must meet the following requirements: Blood routine: Neutrophil count (ANC) ≥ 1.5×10⁹/L; Platelet count (PLT) ≥ 90×10⁹/L; Hemoglobin (Hb) ≥ 90 g/L;Blood biochemistry: Total bilirubin (TBIL) ≤ 2.5×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5×ULN; Alkaline phosphatase ≤ 2.5×ULN; Blood urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5×ULN;
* 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 ms in females (QTcF calculation formula: QTcF = QT/(RR^1/3));
* Voluntarily participate in this study, sign the informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

* Stage IV breast cancer, recurrent or metastatic breast cancer, or inflammatory breast cancer;
* A history of any malignant tumor, or having received anti-tumor treatment or radiotherapy for any malignant tumor in the past, excluding cured malignant tumors such as carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin;
* Concurrent participation in other clinical trials;
* Having received blood transfusion or treatment with colony-stimulating factors, etc. within 2 weeks before enrollment;
* Known history of allergy to the components of the drugs in this protocol;
* History of immunodeficiency, including positive HIV test, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation;
* A history of any heart disease, including: angina pectoris; arrhythmia requiring drug treatment or with clinical significance; myocardial infarction; heart failure; any other heart disease judged by the researcher as unsuitable for participating in this trial;
* Pregnant or lactating female patients;
* Any other conditions that the researcher deems make the subject unsuitable for participating in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
3-years Invasive Disease-Free Survival (iDFS) | 36 months from randomization

SECONDARY OUTCOMES:
Distant Disease-Free Survival (DDFS) | Up to 48 months
Overall Survival (OS) | up to 48 months
Incidence and Severity of Adverse Events | From treatment initiation to 30 days after the last dose, up to approximately 36 months
  According to Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0)
Patient-Reported Outcomes (PROs) | Baseline to end of follow-up (up to 48 months)
  EORTC QLQ-C30 (version 3.0) Quality of Life Questionnaire.
  The scores of each domain in the scale need to be converted into a 0 - 100 scale through standardized calculation:
  Functional domains: Higher scores indicate better functional status. Symptom domains: Higher scores indicate more severe symptoms. Global quality of life: Higher scores indicate a better quality of life.

IPD SHARING:
Plan to Share IPD: No